CLINICAL TRIAL: NCT02473926
Title: Targeting Physical Activity to Improve Cardiovascular Health in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-1080; K23HL118133 (NIH)
Record Dates: First submitted 2015-04-24; First posted 2015-06-17 (Estimated); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Motor Activity; Health Behavior; Diabetes Mellitus, Type 2
Keywords: Physical Activity; Physical Function; Physical Impairment; Sedentary Lifestyle
MeSH Terms: conditions — Motor Activity; Health Behavior; Diabetes Mellitus, Type 2; Sedentary Behavior | interventions — Exercise; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity Program Intervention (Experimental): The intervention seeks to increase physical activity and improve strength by addressing individual , behavioral, and social/environmental factors. Health promotion clinic staff will deliver counseling by phone on a bi-weekly basis - a clinic physician assistant will coordinate with the counselor during in-person clinic visits, teach participants to perform strengthening exercise, and assess for safety concerns associated with type 2 diabetes.
  In addition to behavioral counseling targeting social cognitive theory constructs, counselors will assist participants in the intervention group to set specific goals for physical activity in a paper log and on an electronic FitBit activity tracking device.Health promotion clinic staff will encourage participants to advance goals towards meeting U.S. physical activity guidelines of 150 minutes/week of moderate intensity activity and 2-3 days/week of strength activities.
  Interventions: Behavioral: Physical Activity
- Usual Care Group (Other): Participants in the usual care arm will receive three mailings (Intervention Questionnaires) during the intervention phase. Health promotion clinic staff will mail materials from the Center for Disease Control and Prevention website that address general health aging topics.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Physical Activity — Physical Activity Program Intervention
  Arms: Physical Activity Program Intervention
Behavioral: Questionnaires — Participants in the usual care arm will receive three mailings during the intervention phase.
  Arms: Usual Care Group

SUMMARY:
This study plans to learn more about physical activity and physical function in sedentary older adults with type 2 diabetes.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a randomized controlled trial with 1:1 patient-level randomization to an evidence-based physical activity program intervention versus usual care in sedentary older adults with type 2 diabetes in two primary care clinic sites.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes
* Sedentary individual, performing <20 minutes of physical activity on <3 days/week

Exclusion Criteria:

* Dementia (Folstein Mini-Mental Status Exam <24) or clinical diagnosis
* Excessive fall risk: Can not hold semi-tandem stance for >10 seconds
* Type 2 diabetes-related safety concerns: Prior diabetic foot ulcer, Charcot foot, asymptomatic hypoglycemia
* Severely uncontrolled hypertension (BP >180/100)
* Excessive hearing or visual impairment for counseling
* Limited life expectancy: Active treatment for malignancy
* Performs regular physical activity >20 minutes on >3 days/week

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Huebschmann, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver | Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huebschmann AG, Glasgow RE, Leavitt IM, Chapman K, Rice JD, Lockhart S, Stevens-Lapsley JE, Reusch JEB, Dunn AL, Regensteiner JG. Integrating a physical activity coaching intervention into diabetes care: a mixed-methods evaluation of a pilot pragmatic trial. Transl Behav Med. 2022 May 25;12(4):601-610. doi: 10.1093/tbm/ibac014. PMID 35312788

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 55 people were determined to be eligible for this study, however 5 of them withdrew prior to randomization. This explains the discrepancy between Protocol section (n=55) and Participant Flow Module (n=50).
Groups:
- Physical Activity Program Intervention: The intervention seeks to increase physical activity and improve strength by addressing individual , behavioral, and social/environmental factors. Health promotion clinic staff will deliver counseling by phone on a bi-weekly basis - a clinic physician assistant will coordinate with the counselor during in-person clinic visits, teach participants to perform strengthening exercise, and assess for safety concerns associated with type 2 diabetes.
  In addition to behavioral counseling targeting social cognitive theory constructs, counselors will assist participants in the intervention group to set specific goals for physical activity in a paper log and on an electronic FitBit activity tracking device.Health promotion clinic staff will encourage participants to advance goals towards meeting U.S. physical activity guidelines of 150 minutes/week of moderate intensity activity and 2-3 days/week of strength activities.
  Physical Activity: Physical Activity Program Intervention
Period: Overall Study
Arm/Group | Physical Activity Program Intervention | Usual Care Group
Started | 28 | 22
Completed | 25 | 22
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Activity Program Intervention | Usual Care Group | Total
Number analyzed (Participants) | 28 | 22 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (7.6) | 66.5 (7.1) | 66.5 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 15 | 9 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 26 | 17 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 13 | 12 | 25
  Black/African American | 10 | 4 | 14
  Asian | 2 | 1 | 3
  Alaskan Native/Native American | 1 | 0 | 1
  Hispanic | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 28 | 22 | 50
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 92.0 (21.4) | 90.6 (21.7) | 91.2 (47.0)
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 32.8 (6.0) | 31.6 (6.7) | 32.1 (6.4)
Hemoglobin A1c (%) [Mean (Standard Deviation); unit: percent] | 6.9 (1.3) | 6.7 (0.8) | 6.8 (1.1)
Systolic Blood Pressure (mm/Hg) [Mean (Standard Deviation); unit: mm/Hg] | 128.1 (9.4) | 125.6 (10.5) | 127.0 (9.9)
Diastolic Blood Pressure (mm/Hg) [Mean (Standard Deviation); unit: mm/Hg] | 83.6 (8.6) | 80.0 (8.1) | 82.0 (8.5)
Baseline fitness level (VO2peak, ml/kg/min) [Mean (Standard Deviation); unit: ml/kg/min] | 18.5 (4.7) | 18.3 (3.0) | 18.4 (4.4)
Depressive symptoms by Center for Epidemiologic Studies Depression Scale (CES-D) [Mean (Standard Deviation); unit: points] — Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.
  points | 10.3 (8.3) | 10.2 (8.3) | 10.2 (8.2)
Endurance Confidence Survey [Mean (Standard Deviation); unit: points] — This survey measures confidence in ability to do different things related to physical activity and endurance. The scoring ranges from 0-1,200, with higher scores indicating greater confidence.
  points | 695.0 (372.7) | 584.1 (288.9) | 682.8 (345.8)
Confidence: Motivation to conduct physical activity(PA) amidst competing demands [Mean (Standard Deviation); unit: points] — This survey measures confidence in ability to motivate oneself in order to perform physical activity amidst competing demands. The scoring ranges from 0-60, with higher scores indicating greater confidence.
  points | 41.2 (9.8) | 43.8 (8.6) | 41.7 (11.9)
Confidence: Self-efficacy for physical activity in presence of diabetes [Mean (Standard Deviation); unit: points] — This survey measures confidence in ability to perform physical activity with a type 2 diabetes diagnosis. The scoring ranges from 0-800, with higher scores indicating greater confidence.
  points | 592.1 (158.6) | 587.3 (183.2) | 588.8 (153.2)
% participants with baseline functional impairment [Count of Participants; unit: Participants] — This is the percentage of participants in each group with functional impairment at entry in the study as measured by the short physical performance battery (SPPB) test. Impairment is identified by an SPPB score of <12, with higher values indicating less functional impairment.
  Participants | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Objective Physical Activity at 4 Months
Description: ActiGraph accelerometer measures physical activity objectively as steps/week. These data are presented as the change from baseline values.
Time Frame: Baseline, 4 Months
Measure: Mean (95% Confidence Interval); unit: steps/week
Arm/Group | Physical Activity Program Intervention | Usual Care Group
Number analyzed (Participants) | 25 | 21
steps/week | 3155 [-2169 to 8478] | 1581 [-5183 to 8344]

2. Secondary Outcome: Change From Baseline in Physical Function at 4 Months
Description: Measured via 400-meter rapid gait speed test. These data are presented as the change from baseline values, where decrease in numbers indicate a faster walking speed.
Time Frame: Baseline, 4 Months
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Physical Activity Program Intervention | Usual Care Group
Number analyzed (Participants) | 25 | 22
seconds | -23.4 [-46.5 to -0.3] | 7.3 [-17.6 to 32.3]

3. Secondary Outcome: Change From Baseline in Physical Function at 4 Months
Description: Measured via the Short Physical Performance Battery (SPPB), which evaluates balance, usual walking speed, and repeated chair rise. These data are presented as the change from baseline values where higher values indicate better physical function (scoring range 0-12).
Time Frame: Baseline, 4 Months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Physical Activity Program Intervention | Usual Care Group
Number analyzed (Participants) | 25 | 22
units on a scale | 0.9 [0.1 to 1.8] | -0.1 [-0.6 to 0.4]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Physical Activity Program Intervention | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/22
Other Adverse Events (participants affected / at risk) | 3/28 | 0/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Activity Program Intervention (N=28) | Usual Care Group (N=22)
Unrelated Medical Issue (Psychiatric disorders) | 1 (1) | 0 (0) — Major depressive episode with suicidal ideation
Unrelated Medical Issue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Spinal injury in a motor vehicle accident
Unrelated Medical Issue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — exacerbation of chronic knee arthritis pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT02473926/Prot_SAP_000.pdf